CLINICAL TRIAL: NCT05991245
Title: French National Cohort MATRIX "Renal and Systemic Thrombotic Microangiopathy"
Acronym: MATRIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RNI/MATRIX; F20221110095846 (Registry Identifier: CNIL); 2022-59 (Registry Identifier: Ethique CVL)
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Thrombotic Microangiopathy; Acute Kidney Injury; Hemolytic Uremic Syndrome; Nephrology; Kidney Diseases
Keywords: Thrombotic microangiopathy; Acute kidney injury; Hemolytic uremic syndrome; Kidney histology; Complement
MeSH Terms: conditions — Thrombotic Microangiopathies; Acute Kidney Injury; Hemolytic-Uremic Syndrome; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, Tissue and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MATRIX: Thrombotic microangiopathy with kidney biopsy
  Interventions: Other: Collecting datas

INTERVENTIONS:
Other: Collecting datas — Blood, Tissue and Urine samples

SUMMARY:
Thrombotic microangiopathies (TMAs) are a diverse, rare but serious group of diseases. Progress has been made regarding the epidemiology of TMA (Bayer CJASN 2019). It has been shown that secondary TMAs account for 95% of cases, whereas primary TMAs (atypical hemolytic syndromes (HUS) and thrombotic thrombocytopenic purpura (TTP)) account for only about 5%.

However, in many cases, the pathophysiology, optimal management and prognosis of TMA remains unclear and it has been shown that patients with TMA may have renal-limited TMA or renal and hematological TMA (ie. With (mechanical anemia, thrombocytopenia, elevated LDH, decreased haptoglobin, schistocytes). In most studies, kidney biopsies are not performed and the diagnostic workup is uncomplete.

As this is a rare disease, only a multicenter approach (>20 centers) over a long period of time (>10 years), with adequate diagnostic workup including kidney biopsies can help us to answer these questions (investigators in the present are usually members of the CNR-MAT (a network of the TMA centers in France).

DETAILED DESCRIPTION:
Thrombotic microangiopathies (TMAs) are a diverse, rare but serious group of diseases. Their epidemiology has recently been elucidated thanks to work published by our team. It has been shown that secondary TMAs account for 95% of cases, whereas primary TMAs (atypical hemolytic syndromes (HUS) and thrombotic thrombocytopenic purpura (TTP)) account for only about 5%.

However, many epidemiologic problems remain. First, many but not all patients with TMA as classically defined (mechanical anemia, thrombocytopenia, elevated LDH, decreased haptoglobin, schizocytes) have impaired renal function. If a renal biopsy is performed (which is not always the case, as TMA is a risk factor for bleeding after renal biopsy), the renal lesions do not always show "renal-limited" TMA. We also do not know which of the causes of systemic TMA are associated with renal TMA and which are not.

Conversely, in patients with renal biopsy, we can find stigmata of renal-limited TMA in the absence of systemic TMA. Why do some patients have systemic TMA but not renal TMA and others have renal TMA but not systemic TMA? Most studies are based on a few small clinical cases and the literature reviews that report them.

The vital, renal, and cardiovascular prognosis of patients with TMA obviously depends on the cause, the clinical presentation of the patients, and their management. However, the renal, systemic, and vital outcomes of renal-only vs. systemic-only vs. systemic and renal TMA, regardless of the cause and severity of TMA, are currently unknown.

As this is a rare disease, only a multicenter approach (>20 centers) over a long period of time (>10 years), including highly recruited university and general hospitals, with experienced and motivated investigators, can help us to answer these currently unanswered questions (these investigators usually belong to the competence centers of the national reference center).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age or older
2. Who have undergone renal biopsy of the native kidney for impaired renal function between 2009 and July 2022.
3. Presence of classically defined systemic MAT (most of the following parameters: elevated LDH, decreased haptoglobin, schizocytes, thrombocytopenia and anemia) AND/OR presence of arteriolar or glomerular renal MAT as indicated by the pathologist (including endothelial turgor, mesangiolysis, double contours, presence of thrombi, fibrinoid necrosis of the arterial wall).

Exclusion Criteria:

1. Kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population corresponds to French adult nephrology patients with renal and/or systemic thrombotic microangiopathy, for whom renal biopsy data are available. It is not extendable to renal transplant patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Presence of isolated renal, hematological or renal associated with hematological features ot thrombotic microangiopathies | 1/ Baseline, ie date of kidney biopsy
  Clinical data

SECONDARY OUTCOMES:
Assess correlations between specific anatomopathological lesions and thrombotic microangiopathies phenotypes | 1/ Baseline, ie date of kidney biopsy
  Pathological and clinical data
Assess correlations between cause of thrombotic microangiopathies and clinical phenotypes | 1/ Baseline, ie date of kidney biopsy
  Clinical data
Define the biological profile (standard biology and alternative complement pathway analyses including genetic data) of these thrombotic microangiopathies. | 1/ Up to 2 weeks after baseline date ; 2/ Date of last follow-up, an average of 2 years
  Biological data
Define the renal, cardiovascular and vital prognosis of these patients | 1/ Hospital discharge date, an average of 2 weeks ; 2/ Date of last follow-up, an average of 2 years
  Clinical data
Define treatments for these patients | 1/ Hospital discharge date, an average of 2 weeks
  Clinical data

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Halimi, MD, PhD, Study Director — CHRU TOURS, Nephrology; Valentin Maisons, MD, Principal Investigator — CHRU TOURS, Nephrology
Locations (1):
- Department of Nephrology, University Hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goodship TH, Cook HT, Fakhouri F, Fervenza FC, Fremeaux-Bacchi V, Kavanagh D, Nester CM, Noris M, Pickering MC, Rodriguez de Cordoba S, Roumenina LT, Sethi S, Smith RJ; Conference Participants. Atypical hemolytic uremic syndrome and C3 glomerulopathy: conclusions from a "Kidney Disease: Improving Global Outcomes" (KDIGO) Controversies Conference. Kidney Int. 2017 Mar;91(3):539-551. doi: 10.1016/j.kint.2016.10.005. Epub 2016 Dec 16. PMID 27989322
- [Background] Bayer G, von Tokarski F, Thoreau B, Bauvois A, Barbet C, Cloarec S, Merieau E, Lachot S, Garot D, Bernard L, Gyan E, Perrotin F, Pouplard C, Maillot F, Gatault P, Sautenet B, Rusch E, Buchler M, Vigneau C, Fakhouri F, Halimi JM. Etiology and Outcomes of Thrombotic Microangiopathies. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):557-566. doi: 10.2215/CJN.11470918. Epub 2019 Mar 12. PMID 30862697
- [Background] Genest DS, Patriquin CJ, Licht C, John R, Reich HN. Renal Thrombotic Microangiopathy: A Review. Am J Kidney Dis. 2023 May;81(5):591-605. doi: 10.1053/j.ajkd.2022.10.014. Epub 2022 Dec 10. PMID 36509342
- [Derived] Halimi JM, Duval A, Chardon E, Mesnard L, Frimat M, Fakhouri F, Grange S, Servais A, Cartery C, Coppo P, Titeca-Beauport D, Roger S, Baroukh N, Fage N, Delmas Y, Querard AH, Seret G, Bobot M, Le Quintrec M, Ville S, von Tokarski F, Chauvet S, Wynckel A, Martins M, Schurder J, Barbet C, Sautenet B, Gatault P, Caillard S, Antunes C, Bayer G, Philipponnet C, Audard V, Maillard N, Vuiblet V, Gnemmi V, El Ouafi Z, Canet S, Dekeyser M, Piver E, Maisons V; MATRIX Consortium Group. Diagnostic Value of Biological Parameters in Biopsy-Confirmed Thrombotic Microangiopathy-MATRIX Consortium Group. Kidney Int Rep. 2025 Mar 17;10(6):1950-1959. doi: 10.1016/j.ekir.2025.03.019. eCollection 2025 Jun. PMID 40630316